CLINICAL TRIAL: NCT04570475
Title: High Dose Vitamin D Plus Multivitamin in the Prevention of Cluster Headache: a Randomized, Double-blind, Placebo Controlled Trial.
Brief Title: High Dose Vitamin D Plus Multivitamin in the Prevention of Cluster Headache
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low number met criteria to randomize.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mark J Burish, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-20-0945
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cluster Headache
Keywords: headache; trigeminal autonomic cephalalgia; chronic cluster headache; episodic cluster headache
MeSH Terms: conditions — Cluster Headache; Headache; Trigeminal Autonomic Cephalalgias | interventions — Vitamin D; Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin D+multivitamin (Experimental)
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: multivitamin
- placebo+multivitamin (Active Comparator)
  Interventions: Dietary Supplement: multivitamin; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Participants will receive vitamin D+multivitamin for 3 weeks. At the end of 3 weeks they will complete an online or paper questionnaire and blood work will be done.
  Arms: vitamin D+multivitamin
Dietary Supplement: multivitamin — Participants will receive placebo+multivitamin or vitamin D+multivitamin for 3 weeks. At the end of 3 weeks they will complete an online or paper questionnaire and blood work will be done.
Dietary Supplement: Placebo — Participants will receive placebo+multivitamin for 3 weeks. At the end of 3 weeks they will complete an online or paper questionnaire and blood work will be done.
  Arms: placebo+multivitamin

SUMMARY:
This study intends to investigate the use of high-dose Vitamin D3 plus a multivitamin in the prevention of cluster headache attacks.

Participants can be enrolled anywhere in the United States that has access to one of our participating labs (for blood work - anticipated to be available in most of the USA).

The study may include:

* Screening: Participants may be interviewed, examined, fill out surveys, and get blood testing
* Week 1: baseline period (no added medications - to establish a baseline)
* Weeks 2-4: double-blinded experimental period - participants receive either 1) high-dose Vitamin D3 + multivitamin, or 2) placebo + multivitamin. Participants also fill out a survey and have blood testing.
* Weeks 5-7: open-label period - ALL participants receive high-dose Vitamin D3 + multivitamin. Participants also fill out a survey and may have blood testing.

Specifically, our primary outcome is the change from baseline to experimental weeks 1-3 in the frequency of cluster headache attacks between placebo and high-dose vitamin D. Specific primary and secondary outcomes are listed below.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of episodic cluster headache according to the International Classification of Headache Disorders 3rd edition as well as cluster periods that are predictable and have a duration of 6 weeks or greater and approximately one attack daily minimum OR
* A diagnosis of chronic cluster headache according to the International Classification of Headache Disorders 3rd edition as well as approximately one attack daily
* Participants who are unlikely to need to change their preventive cluster headache treatment regimen in the next 6 weeks.

Exclusion Criteria:

* Co-existing disease or other characteristic that precludes appropriate diagnosis of cluster headache.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator,would interfere with adherence to study requirements.
* Inability or unwillingness of subject to give informed consent.
* Known allergy to study drug, multivitamin, or placebo components
* Pregnancy or lactation (breastfeeding)
* Usage of greater than 4,000 International Units of Vitamin D3 daily within 60 days of the beginning of the study.
* Concurrent use of Vitamin D and/or multivitamin along with the inability to stop them before the study begins.
* Liver failure or known coagulation disorder (as this study includes vitamin K) such as haemophilia, von Willebrand disease, Factor V Leiden, Antithrombin III deficiency, Protein C or S deficiency, or anti-phospholipid antibody syndrome.
* A personal medical history of more than 1 deep venous thrombosis and/or pulmonary embolism (as this study includes vitamin K).
* Current use of anticoagulants (as this study includes vitamin K). Anticoagulants include: apixaban (Eliquis), betrixaban (Bevyxxa), dabigatran (Pradaxa), dalteparin (Fragmin), edoxaban (Savaysa), enoxaparin (Lovenox), fondaparinux (Arixtra), heparin, rivaroxiban (Xarelto), and warfarin (Coumadin).
* Current use of medications that alter vitamin D metabolism, including steroids,interferon, phenytoin, phenobarbital, digitalis/digoxin, and thiazide diuretics (such as hydrochlorothiazide or chlorthalidone)
* Participants who are aware that their most recent labwork in the last 2 years showed any of the following:

  1. 25-hydroxyvitamin D levels >75 nmol/L
  2. Elevated calcium level
  3. Elevated phosphate level
  4. Abnormal parathyroid hormone levels
  5. Elevated creatinine level
  6. Of note if any values are outside the acceptable range for the study, candidates may still participate in the study if the most recent lab testing is inside the acceptable range for the study. For example, if a candididate were taking a vitamin or medication that may have caused these elevated levels, but no longer take the vitamin or medication, they may be enrolled if retesting is normal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Change in average weekly frequency of cluster headache attacks | (baseline, average of weeks 1-3)
  First primary outcome
Change in average weekly frequency of cluster headache attacks | (baseline, week 3)
  Second primary outcome

SECONDARY OUTCOMES:
Number of participants who had a reduction of at least 50% in the weekly frequency of cluster headache attacks between baseline and week 3 | (baseline, week 3)
Number of participants who had a reduction of at least 30% in the weekly frequency of cluster headache attacks between baseline and week 3 | baseline, week 3
Change in number of abortive medications or other treatments used per week | baseline, week 3
Change in intensity of cluster headache attacks as assessed by numerical rating scale | baseline, week 3
  Total score ranges from 0-10, and a higher score indicates a greater intensity of attacks
Change in number of participants whose disease is 'much better' or 'very much better' as assessed by the Patient Global Impression of Improvement Scale | baseline, week 3
  With the Patient Global Impression of Improvement Scale, a patient is asked to rate their disease as Very much better, Much better, A little better, No change, A little worse, Much worse, or Very much worse compared to a reference point in the past
Change in quality of life as measured by the Cluster Headache Quality of life questionnaire | baseline, week 3
  Total score ranges from 0-100, and a higher score indicates a better quality of life
Change in duration of cluster headache attacks, in minutes | baseline, week 3
Change in level of 25-hydroxyvitamin D | baseline, week 3
Change in average weekly frequency of cluster headache attacks | (baseline, week 6)
Number of participants who had a reduction of at least 50% in the weekly frequency of cluster headache attacks between baseline and week 6 | (baseline, week 6)
Number of participants who had a reduction of at least 30% in the weekly frequency of cluster headache attacks between baseline and week 6 | baseline, week 6
Change in number of abortive medications or other treatments used per week | baseline, week 6
Change in intensity of cluster headache attacks as assessed by numerical rating scale | baseline, week 6
  Total score ranges from 0-10, and a higher score indicates a greater intensity of attacks
Change in number of participants whose disease is 'much better' or 'very much better' as assessed by the Patient Global Impression of Improvement Scale | baseline, week 6
  With the Patient Global Impression of Improvement Scale, a patient is asked to rate their disease as Very much better, Much better, A little better, No change, A little worse, Much worse, or Very much worse compared to a reference point in the past
Change in quality of life as measured by the Cluster Headache Quality of life questionnaire | baseline, week 6
  Total score ranges from 0-100, and a higher score indicates a better quality of life
Change in duration of cluster headache attacks, in minutes | baseline, week 6
Change in level of 25-hydroxyvitamin D | baseline, week 6
Number of days until end of the cluster period after the start of treatment (i.e., the time to the end of an episodic cluster cycle) | upto 3 weeks from treatment
Change in average weekly frequency of cluster headache attacks | (baseline, week 2)
Change in average weekly frequency of cluster headache attacks | (baseline, week 1)
Change in intensity of cluster headache attacks as assessed by numerical rating scale | baseline, week 2
  Total score ranges from 0-10, and a higher score indicates a greater intensity of attacks
Change in intensity of cluster headache attacks as assessed by numerical rating scale | baseline, week 1
  Total score ranges from 0-10, and a higher score indicates a greater intensity of attacks
Change in duration of cluster headache attacks, in minutes | baseline, week 2
Change in duration of cluster headache attacks, in minutes | baseline, week 1
Change in number of abortive medications or other treatments used per week | baseline, week 2
Change in number of abortive medications or other treatments used per week | baseline, week 1
Change in quality of life as measured by the Cluster Headache Quality of life questionnaire | baseline, week 2
  Total score ranges from 0-100, and a higher score indicates a better quality of life
Change in quality of life as measured by the Cluster Headache Quality of life questionnaire | baseline, week 1
  Total score ranges from 0-100, and a higher score indicates a better quality of life
Change in level of 25-hydroxyvitamin D | baseline, week 2
Change in level of 25-hydroxyvitamin D | baseline, week 1
Change in level of calcium | baseline, week 3
Change in level of calcium | baseline, week 6
Change in level of calcium | baseline, week 2
Change in level of calcium | baseline, week 1
Change in level of phosphate | baseline, week 3
Change in level of phosphate | baseline, week 6
Change in level of phosphate | baseline, week 1
Change in level of phosphate | baseline, week 2
Change in level of parathyroid hormone | baseline, week 3
Change in level of parathyroid hormone | baseline, week 6
Change in level of parathyroid hormone | baseline, week 1
Change in level of parathyroid hormone | baseline, week 2
Change in level of creatinine | baseline, week 3
Change in level of creatinine | baseline, week 6
Change in level of creatinine | baseline, week 1
Change in level of creatinine | baseline, week 2
Change in number of participants whose disease is 'much better' or 'very much better' as assessed by the Patient Global Impression of Improvement Scale | baseline, week 2
  With the Patient Global Impression of Improvement Scale, a patient is asked to rate their disease as Very much better, Much better, A little better, No change, A little worse, Much worse, or Very much worse compared to a reference point in the past
Change in number of participants whose disease is 'much better' or 'very much better' as assessed by the Patient Global Impression of Improvement Scale | baseline, week 1
  With the Patient Global Impression of Improvement Scale, a patient is asked to rate their disease as Very much better, Much better, A little better, No change, A little worse, Much worse, or Very much worse compared to a reference point in the past

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Burish, MD,PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No